CLINICAL TRIAL: NCT01537978
Title: Use of Interactive Gaming After Spinal Cord Injury
Brief Title: Use of Interactive Gaming for Enhanced Function After Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Beatrice Jenny Kiratli PhD, Director Clinical Research Spinal Cord Injury, VA Palo Alto Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18834
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Paraplegia and Tetraplegia
Keywords: spinal cord injury, video gaming, functional improvement
MeSH Terms: conditions — Paraplegia; Quadriplegia; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Video game play (Experimental): Changes in upper limb; strength, active range of motion, electromyographic activity as well as heart rate response.
  Interventions: Other: Video gaming for enhanced function after spinal cord injury.

INTERVENTIONS:
Other: Video gaming for enhanced function after spinal cord injury. — Spinal cord injured indviduals will play Nintendo Wii sports games for an 8 week period.
  Other Names: Nintendo Wii Video gaming

SUMMARY:
The purpose of this study is to evaluate whether there are functional improvements in arm muscles and movments for spinal cord injured indviduals after performing video gaming.

DETAILED DESCRIPTION:
Today, Nintendo's Wii has become integrated into our popular culture replete with its own vocabulary and marketed promise of achieving fitness through video gaming. Recently the term "Wii-habilitation" has gained popularity to represent application of interactive gaming into the therapeutic setting as a form of rehabilitation. However, this technology remains largely untested in the rehabilitation field despite seemingly widespread use.

Interactive gaming may indeed contribute to an important problem in rehabilitation, especially for persons with spinal cord injury (SCI) who use manual wheelchairs for primary mobility and depend on their upper extremity for independence. Individuals with SCI will benefit tremendously by maximization of early rehabilitation post-injury and effective ongoing conditioning focused on the upper extremity through a continuum of care model that supports life-long health habits. Further, traditional exercise therapy targets components of function such as range of motion and strength, but often relies on isolated movements and repetitions which might not be the most effective method. Alternately, video interactive gaming can provide an engaging, variable, challenging, and fun activity-based approach that could enhance both adherence to exercise and functional outcomes.

A video gaming system can be readily implemented in a clinical setting and affordably deployed for home use with minimal instruction, is easy to use for continuation of therapy, and is well-suited to the SCI population for whom exercise options are limited. A wide variety of activities and games are available that utilize upper extremity movements "playing" real world sports such as golf, tennis, and bowling; multiple options for play are available which add variety and contribute to a comprehensive work-out. Players must grade whole upper limb forces to play the various games paralleling a traditional exercise regimen; visual and auditory feedback add interest and fun to the sessions. Interactive gaming allows for single and multiple player options and thus lends itself readily to promotion of social engagement. Real-life scenarios may contribute to self-motivation.

ELIGIBILITY:
Inclusion Criteria:

Neurologic level of injury at or below cervical level 5 (C5) through C8 [tetraplegia] and at or below T1 through L3 [paraplegia]; persons with incomplete lesions at higher levels may be eligible, decided on a case by case basis depending on functional ability, Complete and incomplete injury allowed, Physical capability (ie, sufficient voluntary motor function) to participate in unassisted resistive exercise, determined as a minimum of grade 3 (by manual muscle testing) on elbow and wrist extension, Use of either a manual or power wheelchair as primary mobility, Absence of significant medical complications, Normal or nearly normal cognitive function (ie, minimal cognitive impairment may be allowed on a case by case basis), Willingness to participate for the duration of the study.

Exclusion Criteria:

Use of ambulation for mobility, Concurrently participating in any other exercise intervention or sports program, Medical condition that would interfere in gaming either short term or during extended play.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Increased Electromyographic actvity of upper the upper arm with video gaming. | Testing session 1 - at the start of the study ("week 0"). This is called the baseline testing session.
  EMG will be measured at baseline testing for video game play and post testing after the videogaming is completed.

SECONDARY OUTCOMES:
Increased heart rate with Video gaming | Testing session 1 - at the start of the study ("week 0"). This is called the baseline testing session.
  Baseline heart rate will be measured across all video games to see whcih elicit elevated hear rates consistent with appropriate exercise response.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice J Kiratli, PhD, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- Va Palo Alto Health Care System, Palo Alto, California, United States